CLINICAL TRIAL: NCT07039045
Title: A Phase 1, Open-label, 2-part Study of the Absorption, Metabolism, Excretion, and Bioavailability of [14C]-LY4065967 in Healthy Male Participants
Brief Title: A Study of [14C]-LY4065967 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 27203; J4X-MC-LWCB (Other: Eli Lilly and Company)
Record Dates: First submitted 2025-06-19; First posted 2025-06-26 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- [14C]-LY4065967 Part 1 (Experimental): A single dose containing [14C]-LY4065967.
  Interventions: Radiation: [14C]-LY4065967 Oral
- LY4065967 Part 2 (Experimental): A single dose of LY4065967 followed by a single dose of [14C]-LY4065967.
  Interventions: Drug: LY4065967; Radiation: [14C]-LY4065967 IV

INTERVENTIONS:
Drug: LY4065967 — Oral dose
  Arms: LY4065967 Part 2
Radiation: [14C]-LY4065967 Oral — Oral dose
  Arms: [14C]-LY4065967 Part 1
Radiation: [14C]-LY4065967 IV — IV dose
  Arms: LY4065967 Part 2

SUMMARY:
The purpose of this study is to investigate the absorption, metabolism, excretion, and bioavailability of LY4065967 in healthy male participants. This is a 2-part study. The study will last about 58 days for participants in Part 1 and about 60 days for participants in Part 2.

ELIGIBILITY:
Inclusion Criteria:

* Are overtly healthy as determined by medical evaluation including medical history, physical examination, laboratory tests, and 12-lead electrocardiograms (ECGs).
* Have clinical laboratory test results within normal reference range for the population or investigative site, or results with acceptable deviations that are judged to be not clinically significant by the investigator.
* Have venous access sufficient to allow for blood sampling.
* Currently have a minimum of 1 bowel movement per day.
* Have a body mass index within 18.0 to 35.0 kg/m², inclusive
* Assigned male at birth

Exclusion Criteria

* Have significant previous or current history of cardiovascular, respiratory, hepatic, renal, GI, endocrine, hematological, neurological, thromboembolism, or bleeding disorder capable of significantly altering the absorption, metabolism, or elimination of drugs; of constituting a risk when taking the study intervention; or of interfering with the interpretation of data.
* Have a significant history of or current psychiatric disorders.
* Have history of stomach or intestinal surgery or resection that would potentially alter absorption or excretion of orally administered drugs. Uncomplicated appendectomy, uncomplicated cholecystectomy, and hernia repair will be allowed.
* Have a history of significant chronic constipation or have had acute constipation within 3 weeks prior to check-in.
* Have any abnormality in the 12-lead ECG at screening that, in the opinion of the investigator, increases the risks associated with participating in the study or may confound ECG analysis.
* Have an abnormal blood pressure or pulse rate as determined by the investigator.
* Have known allergies to LY4065967, related compounds, or any components of the formulation, or history of significant atopy.
* Are currently enrolled in or have participated within the last 3 months in a clinical study involving an investigational product or any other type of medical research judged not to be scientifically or medically compatible with this study. If the previous investigational product has a long t1/2, 5 half-lives or 30 days, whichever is longer, should have passed prior to check-in.
* Have previously completed or withdrawn from this study or any other study investigating LY4065967 and have previously received LY4065967.
* Part 2 only: Total [14C]-radioactivity measured in plasma exceeding 2.5 × the standard biological carbon ratio, 50 pMC when analyzed with carbon carrier radiodilution or 250 pMC when analyzed without carbon carrier dilution.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2025-06-23 (Actual); Primary Completion 2025-08-16 (Actual); Study Completion 2025-08-16 (Actual)

PRIMARY OUTCOMES:
Part 1: Percentage of Total Radioactive Dose in Urine and Fecal Excretion | Baseline through Study Completion (21 days)
Part 2: Plasma Area Under the Concentration-time Curve from Zero to Infinity (AUC(0-ꝏ)) for LY4065967 | Baseline through Study Completion (9 Days)

SECONDARY OUTCOMES:
Part 1 Pharmacokinetic (PK): Plasma AUC(0-ꝏ) for Total Radioactivity and LY4065967 | Baseline through Study Completion (21 days)
Part 1 PK: Plasma Maximum Concentration (Cmax) for Total Radioactivity and LY4065967 | Baseline through Study Completion (21 days)
Part 1 PK: Blood Total Radioactivity AUC | Baseline through Study Completion (21 days)
Part 1 PK: Blood Total Radioactivity Cmax | Baseline through Study Completion (21 days)
Part 1: Total Number and Identification of Metabolites | Baseline through Study Completion (21 days)
Part 2 PK: Plasma AUC(0-ꝏ) for Total Radioactivity, [14C]-LY4065967, and LY4065967 | Baseline through Study Completion (9 Days)
Part 2 PK: Plasma Cmax for Total Radioactivity, [14C]-LY4065967, and LY4065967 | Baseline through Study Completion (9 Days)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- Fortrea Clinical Research Unit, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No